CLINICAL TRIAL: NCT05344222
Title: Effects of Photobiomodulation Conditioning of Orofacial Tissue in Surgery for Removal of Impacted Mandibular Third Molars: Randomized, Sham-controlled, Double-blind Clinical Trial
Brief Title: Effects of Photobiomodulation Conditioning in Impacted Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Clinical professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HALIURO
Record Dates: First submitted 2022-03-31; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: An external investigator was assigned to perform randomization. Containing the type of treatment to be used inside, unidentified envelopes were drawn among the participants, resulting in two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (Experimental): The participants in the active photobiomodulation group will be irradiated with infrared LED at a wavelength of 850 nm perpendicular to the surface of the skin in gentle stationary contact at three extraoral points. Treatment will be administered one hour prior to the surgical procedure as well as 48 hours and seven days (removal of sutures) after the first irradiation.
  Interventions: Device: Infrared LED
- Sham Photobiomodulation (Sham Comparator): For the participants in the sham group, a device with a similar appearance will be used that did not emit radiation. Treatment will be administered one hour prior to the surgical procedure as well as 48 hours and seven days (removal of sutures) after the first irradiation.
  Interventions: Device: Similar device - Infrared ED

INTERVENTIONS:
Device: Infrared LED — The participants in the active photobiomodulation group will be irradiated with infrared LED at a wavelength of 850 nm perpendicular to the surface of the skin in gentle stationary contact at three extraoral points. Treatment will be administered one hour prior to the surgical procedure as well as 48 hours and seven days (removal of sutures) after the first irradiation.
  Arms: Photobiomodulation
Device: Similar device - Infrared ED — For the participants in the sham group, a device with a similar appearance will be used that did not emit radiation. Treatment will be administered one hour prior to the surgical procedure as well as 48 hours and seven days (removal of sutures) after the first irradiation.
  Arms: Sham Photobiomodulation

SUMMARY:
The removal of third molars should be considered to avoid problems such as cysts and other complications. Surgical intervention with the manipulation of oral tissues has the undesirable postoperative effects of pain, trismus (limited mouth opening) and edema. Photobiomodulation has also proved effective regarding reductions in pain, edema and trismus. The aim of the present study was to evaluate the effectiveness of photobiomodulation for the conditioning of tissues involved in the surgical removal of impacted mandibular third molars in terms of reducing or eliminating postoperative pain, trismus and edema.

DETAILED DESCRIPTION:
The investigator will select 62 patients from Nove de Julho Clinics, minimal 18 years old, with impacted third molar teeth. The volunteers will be randomly allocated to two groups using a block randomization process: photobiomodulation group (PG) and sham group (SG). The same surgeon and assistant performed all operations. The surgeon, assistant and patients will be all blinded to the LED treatment protocol. The participants in the active photobiomodulation group will be irradiated with infrared LED at a wavelength of 850 nm 08J 80 seconds perpendicular to the surface of the skin in gentle stationary contact at three extraoral points. For the participants in the sham group, a device with a similar appearance will be used that did not emit radiation. Treatment will be administered one hour prior to the surgical procedure as well as 48 hours and seven days (removal of sutures) after the first irradiation. The visual analog scale will be used for the measurement of pain intensity, facial measurements evaluated edema. Mouth opening range will be measured with sterilized manual calipers between the incisal edge of the maxillary and mandibular central incisors. The distribution of the data (normal or non-normal) will be determined using the Shapiro-Wilks test. Data with normal distribution will be analyzed using two-way repeated-measures analysis of variance (ANOVA), the t-test for two groups with independent measures and the paired t-test for two groups with dependent measures. Data with non-normal distribution will be analyzed using the Wilcoxon test for paired data and the Mann-Whitney test for independent data. Categorical data will be analyzed using Fisher's exact test for independent data and McNemar's test for paired data. The significance level will be set at α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* male and female adults (18 years of age or older)
* no tumors in the oral region,
* not having undergone psychiatric treatment in the previous year,
* good general health,
* satisfactory oral hygiene,
* impacted mandibular third molar
* signed statement of informed consent.

Exclusion Criteria:

* habitual use of analgesic or anti-inflammatory medication for other comorbidities,
* undergoing neurological/psychiatric treatment,
* teeth with lesions to be treated in the same hemi-arch as the tooth to be removed,
* systemic disease,
* current smoking habit,
* pericoronitis in the previous 30 days,
* pregnant or nursing women,
* poor oral hygiene,
* photosensitivity disorder,
* tumor in the oral region,
* heart disease,
* diabetes,
* blood dyscrasia,
* chemical dependency,
* allergy to medications used in the study,
* ankylosis of the temporomandibular joint
* intraoperative complications with surgery time exceeding 90 minutes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Infrared Led. | Throught study completion, an average 48
  In the immediate pre-surgery period, three measurements were taken on the face of the patient with a previously sterilized flexible metric tape (centimeters): tragus - pogonion; tragus - lip commissure; and angle of mandible - outer orbicular commissure. Mouth opening range was measured (centimeters) with sterilized manual calipers between the incisal edge of the maxillary and mandibular central incisors The visual analog scale was used for the measurement of pain intensity. Each patient marked a point along a line between two extremes numbered zero (no pain) to 10 (worst possible pain) to represent the pain felt at moment of evaluation (69,70).
Infrared LED - similar device | Throught study completion, an average 48
  In the immediate pre-surgery period, three measurements were taken on the face of the patient with a previously sterilized flexible metric tape (centimeters): tragus - pogonion; tragus - lip commissure; and angle of mandible - outer orbicular commissure. Mouth opening range was measured (centimeters) with sterilized manual calipers between the incisal edge of the maxillary and mandibular central incisors.
  The visual analog scale was used for the measurement of pain intensity. Each patient marked a point along a line between two extremes numbered zero (absence of pain) to 10 (worst pain imaginable) to represent the pain felt at moment of evaluation (69,70).

CONTACTS AND LOCATIONS:
Overall Officials: ERIKA MELLO, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho (UNINOVE), São Paulo, Brazil

REFERENCES:
- [Result] Selimovic E, Ibrahimagic-Seper L, Sisic I, Sivic S, Huseinagic S. Prevention of trismus with different pharmacological therapies after surgical extraction of impacted mandibular third molar. Med Glas (Zenica). 2017 Feb 1;14(1):145-151. doi: 10.17392/871-16. PMID 27612525
- [Result] Lopez-Ramirez M, Vilchez-Perez MA, Gargallo-Albiol J, Arnabat-Dominguez J, Gay-Escoda C. Efficacy of low-level laser therapy in the management of pain, facial swelling, and postoperative trismus after a lower third molar extraction. A preliminary study. Lasers Med Sci. 2012 May;27(3):559-66. doi: 10.1007/s10103-011-0936-8. Epub 2011 May 27. PMID 21617973
- [Result] Kocer G, Yuce E, Tuzuner Oncul A, Dereci O, Koskan O. Effect of the route of administration of methylprednisolone on oedema and trismus in impacted lower third molar surgery. Int J Oral Maxillofac Surg. 2014 May;43(5):639-43. doi: 10.1016/j.ijom.2013.11.005. Epub 2013 Dec 12. PMID 24332587
- [Result] Fernandes IA, de Souza GM, Pinheiro MLP, Falci SGM. Intramuscular injection of dexamethasone for the control of pain, swelling, and trismus after third molar surgery: a systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2019 May;48(5):659-668. doi: 10.1016/j.ijom.2018.09.014. Epub 2018 Oct 14. PMID 30327153
- [Result] Leal Junior EC, Lopes-Martins RA, Frigo L, De Marchi T, Rossi RP, de Godoi V, Tomazoni SS, Silva DP, Basso M, Filho PL, de Valls Corsetti F, Iversen VV, Bjordal JM. Effects of low-level laser therapy (LLLT) in the development of exercise-induced skeletal muscle fatigue and changes in biochemical markers related to postexercise recovery. J Orthop Sports Phys Ther. 2010 Aug;40(8):524-32. doi: 10.2519/jospt.2010.3294. PMID 20436237
- [Result] Toma RL, Tucci HT, Antunes HK, Pedroni CR, de Oliveira AS, Buck I, Ferreira PD, Vassao PG, Renno AC. Effect of 808 nm low-level laser therapy in exercise-induced skeletal muscle fatigue in elderly women. Lasers Med Sci. 2013 Sep;28(5):1375-82. doi: 10.1007/s10103-012-1246-5. Epub 2013 Jan 8. PMID 23296713
- [Result] Vanin AA, Miranda EF, Machado CS, de Paiva PR, Albuquerque-Pontes GM, Casalechi HL, de Carvalho PT, Leal-Junior EC. Erratum to: What is the best moment to apply phototherapy when associated to a strength training program? A randomized, double-blinded, placebo-controlled trial. Lasers Med Sci. 2017 Jan;32(1):253. doi: 10.1007/s10103-016-2121-6. No abstract available. PMID 27924418
- [Result] Ferraresi C, Huang YY, Hamblin MR. Photobiomodulation in human muscle tissue: an advantage in sports performance? J Biophotonics. 2016 Dec;9(11-12):1273-1299. doi: 10.1002/jbio.201600176. Epub 2016 Nov 22. PMID 27874264
- [Result] Leal Junior EC, Lopes-Martins RA, Rossi RP, De Marchi T, Baroni BM, de Godoi V, Marcos RL, Ramos L, Bjordal JM. Effect of cluster multi-diode light emitting diode therapy (LEDT) on exercise-induced skeletal muscle fatigue and skeletal muscle recovery in humans. Lasers Surg Med. 2009 Oct;41(8):572-7. doi: 10.1002/lsm.20810. PMID 19731300
- [Result] Leal Junior EC, Lopes-Martins RA, Baroni BM, De Marchi T, Rossi RP, Grosselli D, Generosi RA, de Godoi V, Basso M, Mancalossi JL, Bjordal JM. Comparison between single-diode low-level laser therapy (LLLT) and LED multi-diode (cluster) therapy (LEDT) applications before high-intensity exercise. Photomed Laser Surg. 2009 Aug;27(4):617-23. doi: 10.1089/pho.2008.2350. PMID 19302015
- [Result] Gautam AP, Fernandes DJ, Vidyasagar MS, Maiya AG, Guddattu V. Low level laser therapy against radiation induced oral mucositis in elderly head and neck cancer patients-a randomized placebo controlled trial. J Photochem Photobiol B. 2015 Mar;144:51-6. doi: 10.1016/j.jphotobiol.2015.01.011. Epub 2015 Feb 7. PMID 25704314
- [Result] Guedes CDCFV, de Freitas Filho SAJ, de Faria PR, Loyola AM, Sabino-Silva R, Cardoso SV. Variation of Energy in Photobiomodulation for the Control of Radiotherapy-Induced Oral Mucositis: A Clinical Study in Head and Neck Cancer Patients. Int J Dent. 2018 Feb 22;2018:4579279. doi: 10.1155/2018/4579279. eCollection 2018. PMID 29681940
- [Result] Marin-Conde F, Castellanos-Cosano L, Pachon-Ibanez J, Serrera-Figallo MA, Gutierrez-Perez JL, Torres-Lagares D. Photobiomodulation with low-level laser therapy reduces oral mucositis caused by head and neck radio-chemotherapy: prospective randomized controlled trial. Int J Oral Maxillofac Surg. 2019 Jul;48(7):917-923. doi: 10.1016/j.ijom.2018.12.006. Epub 2018 Dec 24. PMID 30591391
- [Result] Rezk-Allah SS, Abd Elshaf HM, Farid RJ, Hassan MAE, Alsirafy SA. Effect of Low-Level Laser Therapy in Treatment of Chemotherapy Induced Oral Mucositis. J Lasers Med Sci. 2019 Spring;10(2):125-130. doi: 10.15171/jlms.2019.20. Epub 2019 Feb 25. PMID 31360381
- [Result] Gonzalez-Arriagada WA, Ramos LMA, Andrade MAC, Lopes MA. Efficacy of low-level laser therapy as an auxiliary tool for management of acute side effects of head and neck radiotherapy. J Cosmet Laser Ther. 2018 Apr;20(2):117-122. doi: 10.1080/14764172.2017.1376097. Epub 2017 Dec 4. PMID 29020483
- [Result] Silva LC, Sacono NT, Freire Mdo C, Costa LR, Batista AC, Silva GB. The Impact of Low-Level Laser Therapy on Oral Mucositis and Quality of Life in Patients Undergoing Hematopoietic Stem Cell Transplantation Using the Oral Health Impact Profile and the Functional Assessment of Cancer Therapy-Bone Marrow Transplantation Questionnaires. Photomed Laser Surg. 2015 Jul;33(7):357-63. doi: 10.1089/pho.2015.3911. PMID 26154723
- [Result] Gouvea de Lima A, Villar RC, de Castro G Jr, Antequera R, Gil E, Rosalmeida MC, Federico MH, Snitcovsky IM. Oral mucositis prevention by low-level laser therapy in head-and-neck cancer patients undergoing concurrent chemoradiotherapy: a phase III randomized study. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):270-5. doi: 10.1016/j.ijrobp.2010.10.012. Epub 2010 Dec 14. PMID 21163585
- [Result] Sales PHDH, Barros AWP, Silva PGB, Vescovi P, Leao JC. Is the Er: YAG Laser Effective in Reducing Pain, Edema, and Trismus After Removal of Impacted Mandibular Third Molars? A Meta-Analysis. J Oral Maxillofac Surg. 2022 Mar;80(3):501-516. doi: 10.1016/j.joms.2021.10.006. Epub 2021 Oct 20. PMID 34793714
- [Result] Oguz O. The proportion of the face in younger adults using the thumb rule of Leonardo da Vinci. Surg Radiol Anat. 1996;18(2):111-4. doi: 10.1007/BF01795228. PMID 8782316
- [Result] Rodrigues ED, Pereira GS, Vasconcelos BC, Ribeiro RC. Effect of preemptive dexamethasone and etoricoxib on postoperative period following impacted third molar surgery - a randomized clinical trial. Med Oral Patol Oral Cir Bucal. 2019 Nov 1;24(6):e746-e751. doi: 10.4317/medoral.23095. PMID 31655834
- [Result] Shugars DA, Benson K, White RP Jr, Simpson KN, Bader JD. Developing a measure of patient perceptions of short-term outcomes of third molar surgery. J Oral Maxillofac Surg. 1996 Dec;54(12):1402-8. doi: 10.1016/s0278-2391(96)90253-0. PMID 8957118
- [Result] Braimah RO, Ndukwe KC, Owotade FJ, Aregbesola SB. Oral health related quality of life (OHRQoL) following third molar surgery in Sub-Saharan Africans: an observational study. Pan Afr Med J. 2016 Oct 19;25:97. doi: 10.11604/pamj.2016.25.97.7656. eCollection 2016. PMID 28292060
- [Result] Ibikunle AA, Adeyemo WL. Oral health-related quality of life following third molar surgery with or without application of ice pack therapy. Oral Maxillofac Surg. 2016 Sep;20(3):239-47. doi: 10.1007/s10006-016-0558-1. Epub 2016 May 3. PMID 27139019
- [Result] Cassetta M, Altieri F. The influence of mandibular third molar germectomy on the treatment time of impacted mandibular second molars using brass wire: a prospective clinical pilot study. Int J Oral Maxillofac Surg. 2017 Jul;46(7):905-911. doi: 10.1016/j.ijom.2017.03.027. Epub 2017 Apr 10. PMID 28408148
- [Result] Duarte-Rodrigues L, Miranda EFP, Souza TO, de Paiva HN, Falci SGM, Galvao EL. Third molar removal and its impact on quality of life: systematic review and meta-analysis. Qual Life Res. 2018 Oct;27(10):2477-2489. doi: 10.1007/s11136-018-1889-1. Epub 2018 May 24. PMID 29797177
- [Result] Momeni E, Barati H, Arbabi MR, Jalali B, Moosavi MS. Low-level laser therapy using laser diode 940 nm in the mandibular impacted third molar surgery: double-blind randomized clinical trial. BMC Oral Health. 2021 Feb 18;21(1):77. doi: 10.1186/s12903-021-01434-1. PMID 33602198
- [Result] Asutay F, Ozcan-Kucuk A, Alan H, Koparal M. Three-dimensional evaluation of the effect of low-level laser therapy on facial swelling after lower third molar surgery: A randomized, placebo-controlled study. Niger J Clin Pract. 2018 Sep;21(9):1107-1113. doi: 10.4103/njcp.njcp_38_18. PMID 30156193
- [Result] Alan H, Yolcu U, Koparal M, Ozgur C, Ozturk SA, Malkoc S. Evaluation of the effects of the low-level laser therapy on swelling, pain, and trismus after removal of impacted lower third molar. Head Face Med. 2016 Jul 26;12(1):25. doi: 10.1186/s13005-016-0121-1. PMID 27457369
- [Result] Koparal M, Kucuk AO, Alan H, Asutay F, Avci M. Effects of low-level laser therapy following surgical extraction of the lower third molar with objective measurement of swelling using a three-dimensional system. Exp Ther Med. 2018 Apr;15(4):3820-3826. doi: 10.3892/etm.2018.5921. Epub 2018 Mar 2. PMID 29581740
- [Result] Singh T, More V, Fatima U, Karpe T, Aleem MA, Prameela J. Effect of proteolytic enzyme bromelain on pain and swelling after removal of third molars. J Int Soc Prev Community Dent. 2016 Dec;6(Suppl 3):S197-S204. doi: 10.4103/2231-0762.197192. PMID 28217537
- [Result] Demirsoy MS, Tumer MK, Erdil A, Ozkan Y. Evaluation of the effects of the surgical removal of impacted third molars on the emotional state of individuals with Beck depression inventory. Niger J Clin Pract. 2020 Oct;23(10):1407-1413. doi: 10.4103/njcp.njcp_603_19. PMID 33047698
- [Result] Isolan C, Kinalski MD, Leao OA, Post LK, Isolan TM, Dos Santos MB. Photobiomodulation therapy reduces postoperative pain after third molar extractions: A randomized clinical trial. Med Oral Patol Oral Cir Bucal. 2021 May 1;26(3):e341-e348. doi: 10.4317/medoral.24228. PMID 33340081
- [Result] Uslu MO, Akgul S. Evaluation of the effects of photobiomodulation therapy and ozone applications after gingivectomy and gingivoplasty on postoperative pain and patients' oral health-related quality of life. Lasers Med Sci. 2020 Sep;35(7):1637-1647. doi: 10.1007/s10103-020-03037-8. Epub 2020 May 20. PMID 32435906
- [Result] Eshghpour M, Ahrari F, Takallu M. Is Low-Level Laser Therapy Effective in the Management of Pain and Swelling After Mandibular Third Molar Surgery? J Oral Maxillofac Surg. 2016 Jul;74(7):1322.e1-8. doi: 10.1016/j.joms.2016.02.030. Epub 2016 Mar 12. PMID 27055228
- [Result] Raiesian S, Khani M, Khiabani K, Hemmati E, Pouretezad M. Assessment of Low-Level Laser Therapy Effects After Extraction of Impacted Lower Third Molar Surgery. J Lasers Med Sci. 2017 Winter;8(1):42-45. doi: 10.15171/jlms.2017.08. Epub 2017 Jan 8. PMID 28912943
- [Result] Gil MLB, Marinho LMRF, de Moraes M, Wada RS, Groppo FC, Sato JE, de Sousa MLR. Effectiveness of Acupuncture in Dental Surgery: A Randomized, Crossover, Controlled Trial. J Acupunct Meridian Stud. 2020 Jun;13(3):104-109. doi: 10.1016/j.jams.2020.03.063. Epub 2020 Mar 20. PMID 32205274
- [Result] Domah F, Shah R, Nurmatov UB, Tagiyeva N. The Use of Low-Level Laser Therapy to Reduce Postoperative Morbidity After Third Molar Surgery: A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2021 Feb;79(2):313.e1-313.e19. doi: 10.1016/j.joms.2020.09.018. Epub 2020 Sep 17. PMID 33058775
- [Result] Dawdy J, Halladay J, Carrasco-Labra A, Araya I, Yanine N, Brignardello-Petersen R. Efficacy of adjuvant laser therapy in reducing postsurgical complications after the removal of impacted mandibular third molars: A systematic review update and meta-analysis. J Am Dent Assoc. 2017 Dec;148(12):887-902.e4. doi: 10.1016/j.adaj.2017.06.043. Epub 2017 Oct 5. PMID 28987483
- [Result] Hamid MA. Low-level Laser Therapy on Postoperative Pain after Mandibular Third Molar Surgery. Ann Maxillofac Surg. 2017 Jul-Dec;7(2):207-216. doi: 10.4103/ams.ams_5_17. PMID 29264287
- [Result] Petrini M, Ferrante M, Trentini P, Perfetti G, Spoto G. Effect of pre-operatory low-level laser therapy on pain, swelling, and trismus associated with third-molar surgery. Med Oral Patol Oral Cir Bucal. 2017 Jul 1;22(4):e467-e472. doi: 10.4317/medoral.21398. PMID 28578368
- [Result] Fernandes IA, Armond ACV, Falci SGM. The Effectiveness of the Cold Therapy (cryotherapy) in the Management of Inflammatory Parameters after Removal of Mandibular Third Molars: A Meta-Analysis. Int Arch Otorhinolaryngol. 2019 Apr;23(2):221-228. doi: 10.1055/s-0039-1677755. Epub 2019 Mar 13. PMID 30956709
- [Result] Noba C, Mello-Moura ACV, Gimenez T, Tedesco TK, Moura-Netto C. Laser for bone healing after oral surgery: systematic review. Lasers Med Sci. 2018 Apr;33(3):667-674. doi: 10.1007/s10103-017-2400-x. Epub 2017 Dec 1. PMID 29196831
- [Result] Khorshidi Khiavi R, Pourallahverdi M, Pourallahverdi A, Ghorani Khiavi S, Ghertasi Oskouei S, Mokhtari H. Pain control following impacted third molar surgery with bupivacaine irrigation of tooth socket: a prospective study. J Dent Res Dent Clin Dent Prospects. 2010 Fall;4(4):105-9. doi: 10.5681/joddd.2010.027. Epub 2010 Dec 21. PMID 23346335
- [Result] Sortino F, Cicciu M. Strategies used to inhibit postoperative swelling following removal of impacted lower third molar. Dent Res J (Isfahan). 2011 Oct;8(4):162-71. doi: 10.4103/1735-3327.86031. PMID 22135686
- [Result] de Almeida P, Lopes-Martins RA, Tomazoni SS, Silva JA Jr, de Carvalho Pde T, Bjordal JM, Leal Junior EC. Low-level laser therapy improves skeletal muscle performance, decreases skeletal muscle damage and modulates mRNA expression of COX-1 and COX-2 in a dose-dependent manner. Photochem Photobiol. 2011 Sep-Oct;87(5):1159-63. doi: 10.1111/j.1751-1097.2011.00968.x. Epub 2011 Aug 17. PMID 21749398
- See also: Roochi MM, Heidar H, Kordi S, Bahrami N. Efficacy of low level laser for prevention of pain and trismus after impacted mandibular third molar surgery. J Craniomaxillofacial Res. Published online May 16, 2017:284-288. Accessed January 21, 2021 — https://jcr.tums.ac.ir/index.php/jcr/article/view/141
- See also: Martins M, Garcia MAPY, Fernandes MV, et al. Principais complicações clínicas odontológicas pós-operatórias da cirurgia de terceiro molar incluso/impactado. ConScientiae Saúde. 2010;9(2):278-284 — https://doi.org/10.5585/conssaude.v9i2.2056
- See also: Hummig W, Grossmann E. Use of viminol in acute pain management after third molars extraction. Case report. BrJP. 2018;1(2):188-191. — http://dx.doi.org/10.5935/2595-0118.20180037
- See also: Vicente Â, Loffi AOB, Nesi H. Uso de corticosteroide no pré-operatório em cirurgia de terceiros molares. Rev Bras Odontol. 2013;70(1):22-27. — http://revodonto.bvsalud.org/scielo.php?script=sci_arttext&pid=S0034-72722013000100006
- See also: Medeiros ACR, Branco GLC, Moura LA de. LASER THERAPY IN MOLARS SURGERY IMPACTED: SYSTEMATIC REVIEW. Focus Oral Res. 2019;2(1):59-66. doi:10.35169/for.v2i1.44 — https://doi.org/10.1590/1981-863720170001000023084
- See also: D'Avila RP. Avaliação longitudinal dos efeitos da fototerapia com laser de baixa potência nos movimentos mandibulares, dor e edema após cirurgia ortognática. text. Universidade de São Paulo; 2016 — https://teses.usp.br/teses/disponiveis/23/23149/tde-06032017-120629/pt-br.php
- See also: Ferreira TRR. Drenagem Linfática Manual No Pós-Operatório de Enxerto Ósseo Alveolar: Uma Nova Abordagem Para a Redução Do Edema Facial. PhD Thesis. Universidade de São Paulo; 2010 — https://www.teses.usp.br/teses/disponiveis/61/61132/tde-29072010-104318/pt-br.php
- See also: Gonçalves RD. Abordagem fisioterapêutica no tratamento dos edemas pós cirurgias plásticas. Published online June 12, 2015. Accessed October 25, 2020 — http://dspace.bc.uepb.edu.br/jspui/handle/123456789/10860
- See also: Roochi MM, Heidar H, Kordi S, Bahrami N. Efficacy of low level laser for prevention of pain and trismus after impacted mandibular third molar surgery. J Craniomaxillofacial Res. Published online May 16, 2017:284-288. Accessed January 21, 2021. — https://jcr.tums.ac.ir/index.php/jcr/article/view/141
- See also: Tortorici S, Messina P, Scardina GA, Difalco P. EBSCOhost | 141589931 | EFICÁCIA DA TERAPIA COM LASER DE BAIXO NÍVEL NA INTENSIDADE DA DOR APÓS A EXTRAÇÃO DO TERCEIRO MOLAR INFERIOR. Published 2019. Accessed January 20, 2021. — https://rnp-primo.hosted.exlibrisgroup.com/permalink/f/vsvpiv/TN_cdi_proquest_journals_2415521521
- See also: Peixoto RF, Santos DH, Menezes DP, Araújo D de, Peixoto DF, Silva JS. Controle da dor pós-operatória em cirurgia oral: revisão de literatura. Rev Bras Ciênc Saúde. 2011;15(4):465-470. — https://pesquisa.bvsalud.org/portal/resource/pt/lil-790500
- See also: Effect of 830 nm low-level laser therapy in exercise-induced skeletal muscle fatigue in humans | SpringerLink. Accessed October 28, 2020 — https://link.springer.com/article/10.1007%2Fs10103-008-0592-9
- See also: BDTDUFTM: Influência da laserterapia no desempenho, recuperação e no estresse oxidativo de corredores amadores. Accessed October 28, 2020 — http://bdtd.uftm.edu.br/handle/tede/695
- See also: Miranda SS, Queiroz LR, Freitas VS. PREVENÇÃO E TRATAMENTO DAS MUCOSITES ORAIS: UMA REVISÃO SISTEMÁTICA. Rev Saúde Coletiva UEFS. 2017;6(2):66-73. — https://doi.org/10.13102/rscdauefs.v6i2.1189
- See also: Vannucci MG, Fritzen TN, de Moraes JFD, et al. Estudo comparativo da variabilidade da posição dos terceiros molares retidos em pacientes adolescentes e adultos jovens. Stomatos. 2010;16(31):4-13. — http://revodonto.bvsalud.org/scielo.php?script=sci_abstract&pid=S1519-44422010000200002&lng=es&nrm=iso&tlng=pt
- See also: dos SantosI DR, QuesadaII GAT. Prevalência de terceiros molares e suas respectivas posições se-gundo as classificações de Winter e de Pell e Gregory. Rev Cir Traum Bucomaxilofac. 2009;9(1):83-92. — https://pesquisa.bvsalud.org/portal/resource/pt/lil-524679
- See also: Pereira CB. Informações adicionais sobre o Plano de Frankfurt. Rev AcBO-ISSN 2316-7262. 2013;2(1). — https://silo.tips/download/imagens-na-odontologia-consideraoes-parciais#embed
- See also: Leonardo da Vinci: anatomist | British Journal of General Practice. Accessed October 28, 2020. — https://bjgp.org/content/62/599/319.short
- See also: Markovics ER, Jánosi K, Biriș C, et al. Aesthetic Principles of the Upper Front Teeth: Application of Golden Proportion (Levin) and Golden Percentage (Snow). Acta Marisiensis - Ser Medica. 2013;59(1):25-27 — http://dx.doi.org/10.2478/amma-2013-0005
- See also: Pillon F. Les corticoïdes. Actual Pharm. 2011;50(503):14-21 — https://www.infona.pl/resource/bwmeta1.element.elsevier-456df1cb-a961-37d3-a414-724223fba3f3
- See also: Intan AD, Murdana N, Nuhonni SA, Dwi L, Shatri H. Effect of low-level laser therapy (LLLT) on post-operative pain, trismus and quality of life (QOL) of patients undergoing extraction of impacted lower third molars. J Phys Conf Ser. 2018;1073:042026. — http://dx.doi.org/10.1088/1742-6596/1073/4/042026
- See also: Peimani A, Sardari F, Sarafi S, Sarafi S, Aghdam H, Chiniforush N. The evaluation of photobiomodulation by 980 nm diode laser on postoperative complications after third molar surgery. J Regen Reconstr Restor Triple R. 2018;3(2):x-x. — https://doi.org/10.22037/rrr.v3i2.23050
- See also: Lacerda ÉP de M. Avaliação dos protocolos de crioterapia e termoterapia na morbidade pós cirurgia de terceiros molares inclusos : revisão sistemática e metanálise. Published February 25, 2019. Accessed January 19, 2021 — https://repositorio.ufpe.br/handle/123456789/34114
- See also: Junior N, Do EM. Eficácia da crioterapia na redução da dor, edema e trismo após cirurgia de terceiros molares : revisão sistemática e meta-análise de ensaios clínicos randomizados. Published online January 25, 2019. Accessed January 19, 2021. — http://ri.ufs.br/jspui/handle/riufs/13160
- See also: https://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S0213-12852018000200005 — https://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S0213-12852018000200005
- See also: Sierra SO. Efeito do laser em baixa intensidade sobre a modulação do processo inflamatório pós-cirúrgico: estudo clínico controlado randomizado. — http://bibliotecatede.uninove.br/handle/tede/1031
- See also: Qualidade de vida de pacientes submetidos à exodontia de terceiros molares. Periodikos. Accessed January 22, 2021. — https://www.scielo.br/j/rounesp/a/Q3q5WQKRXcDm3STjD7NV6YG/?format=pdf&lang=pt